CLINICAL TRIAL: NCT04724226
Title: Cryoablation Combined With Camrelizumab and Apatinib
Brief Title: Cryoablation Combined With Camrelizumab and Apatinib in Advanced Hepatocellular Carcinoma
Acronym: C-couple
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fei Gao, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-couple
Record Dates: First submitted 2021-01-25; First posted 2021-01-26 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Cryoablation; Camrelizumab; Apatinib; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; apatinib; Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-couple (Experimental): Camrelizumab and Apatinib after Cryoablation
  Interventions: Drug: Camrelizumab; Apatinib

INTERVENTIONS:
Drug: Camrelizumab; Apatinib — Cryoablation
  Drug: Camrelizumab and Apatinib Camrelizumab (200mg), iv, Q3W; Apatinib (250mg), po, QD
  Other Names: Cryoablation

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of cryoablation combined with pd-1 antibody immunotherapy (Camrelizumab) and anti-angiogenesis therapy (Apatinib) in patients with advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This is a prospective, single arm, phase 2 study to evaluate the efficacy and safety of cryoablation combined with Camrelizumab and Apatinib (C-couple Therapy) in patients with advanced HCC. Subjects who meet the admission criteria will be treated with Camrelizumab and Apatinib after cryoablation until disease progression, intolerable toxicity, death, withdrawal of the patient or the researchers determined that the drug must be discontinued.

The primary outcome measure is to evaluate the objective response rate (ORR) of C-couple Therapy for advanced HCC (BCLC C-stage). The secondary outcome measures include the duration of response (DOR), disease control rate (DCR), progression-free survival rate (PFSR) in 6- and 12-months, overall survival rate (OSR) in 6- and 12-months, the median progression-free survival time (mPFS) and median overall survival time (mOS) of C-couple Therapy for advanced HCC. This study also aims to assess the safety and adverse reactions of C-couple Therapy for advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily joined the study and signed an informed consent form;
2. ≥18 and ≤70 years old, both male and female;
3. Clinically diagnosed or pathologically confirmed advanced hepatocellular carcinoma (unresectable or metastatic), at least one measurable focus without local treatment (according to mRECIST requirements, the measurable focus spiral CT scan length ≥ 10 mm or enlargement Short diameter of lymph node ≥15 mm);
4. Child-Pugh score ≤ 6 points (Child-Pugh A);
5. BCLC staging is stage C; PVTT classification is combined with PVTT (program classification PVTT ≤ 3), and a single lesion in the liver (or multiple lesions with diameter) ≤ 7cm of primary liver cancer.
6. Newly diagnosed patients who have not received targeted therapy or immunotherapy in the past;
7. Able to swallow pills normally;
8. ECOG score: 0～1 (see Annex 1 for ECOG scoring criteria);
9. Expected survival period ≥ 12 weeks;
10. The functions of vital organs meet the following requirements (no blood components, cell growth factors and other corrective treatment drugs are allowed within 14 days before the first administration):

    The absolute count of neutrophils≥1.5×109/L; Platelet ≥80×109/L; Hemoglobin ≥90 g/L; Serum albumin ≥28 g/L; Thyroid-stimulating hormone (TSH)≤1×ULN (if abnormal, the levels of FT3 and FT4 should be examined at the same time, if the levels of FT3 and FT4 are normal, they can be included in the group); Bilirubin≤1.5×ULN (within 7 days before the first administration); ALT and AST ≤3×ULN (within 7 days before the first dose); AKP≤ 2.5×ULN; Serum creatinine≤1.5×ULN;
11. Non-surgical sterilization or female patients of childbearing age need to use a medically approved contraceptive method (such as intrauterine device, contraceptive or condom) during the study treatment period and within 3 months after the end of the study treatment period; Female patients of childbearing age who undergo surgical sterilization must be negative in serum or urine HCG within 72 hours before enrollment in the study; and must be non-lactating; for male patients whose partners are women of childbearing age, Carelil should be given during the trial and at the last time Use effective methods for contraception within 3 months after the onslumab.

Exclusion Criteria:

1. The patient has any active autoimmune disease or a history of autoimmune disease;
2. The patient is using immunosuppressive agents or systemic hormone therapy to achieve the purpose of immunosuppression (dose>10mg/day prednisone or other curative hormones), and continues to use it within 2 weeks before enrollment;
3. The number of system treatment lines ≥ 2 lines;
4. Severe allergic reaction to other monoclonal antibodies;
5. Those with a known history of central nervous system metastasis or hepatic encephalopathy;
6. Patients whose liver tumor burden is greater than 50% of the total liver volume, or who have received liver transplantation in the past;
7. Ascites with clinical symptoms, those who need puncture, drainage, or those who have received ascites drainage within the past 3 months, except those who have only a small amount of ascites on imaging but not accompanied by clinical symptoms;
8. Suffer from high blood pressure and cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
9. Uncontrolled cardiac clinical symptoms or diseases, such as: NYHA level 2 or higher heart failure, unstable angina pectoris, myocardial infarction occurred within 1 year, clinically significant supraventricular or ventricular arrhythmia requires treatment or intervention , QTc>450ms (male); QTc>470ms (female);
10. Abnormal coagulation function (INR>2.0, PT>16s), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy, and allow the preventive use of low-dose aspirin and low molecular heparin;
11. Significant clinically significant bleeding symptoms or clear bleeding tendency occurred within 3 months before randomization, such as pertussis/hemoptysis 2.5ml or more, gastrointestinal bleeding, esophageal and gastric varices with bleeding risk, hemorrhagic stomach Ulcer or vasculitis, etc., if the stool occult blood is positive at the baseline, it can be re-examined. If it is still positive after the re-examination, a gastroscopy is required. If the gastroscope shows severe esophageal and gastric varices, it cannot be included in the group (3 before the group) Except those who have undergone gastroscopy within a month or less to exclude such cases);
12. Arterial/venous thrombosis events that occurred within 6 months before randomization, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
13. Known genetic or acquired bleeding and thrombotic tendency (such as hemophilia patients, coagulation dysfunction, thrombocytopenia, etc.);
14. Urine routine test showed urine protein ≥ ++ and confirmed 24-hour urine protein content> 1.0 g;
15. Patients who have previously received radiotherapy, chemotherapy, hormone therapy, and surgery, after the completion of the treatment (last medication) and less than 4 weeks before the study medication; molecular targeted therapy (including other oral targeted drugs used in clinical trials) is less than the first study medication <5 drug half-lives, or patients whose adverse events (except alopecia) caused by previous treatment have not recovered to ≤ CTCAE level 1;
16. The patient has active infection, fever of unknown origin within 7 days before medication ≥38.5℃, or baseline white blood cell count >15×109/L;
17. Patients with congenital or acquired immune deficiencies (such as HIV-infected persons);
18. Patients with HBV DNA>2000 IU/ml (or 104 copies/ml), HCV RNA>103 copies/ml, HBsAg+ and anti-HCV antibody positive;
19. The patient suffered from other malignant tumors in the past 3 years or at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ);
20. Patients with bone metastases who received palliative radiotherapy within 4 weeks before participating in the study >5% of the bone marrow area;
21. The patient has previously received other anti-PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1, or has previously received apatinib therapy;
22. Live vaccine may be vaccinated less than 4 weeks before study medication or may be administered during the study period;
23. According to the judgment of the investigator, the patient has other factors that may affect the results of the study or cause the study to be terminated halfway, such as alcoholism, drug abuse, other serious diseases (including mental illness) that require combined treatment, and serious laboratory tests Abnormalities, accompanied by family or social factors, will affect the safety of patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 and mRECIST | From date of first dose of study drug until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to 2 years)
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1 and mRECIST

SECONDARY OUTCOMES:
Disease control rate (DCR) | From date of first dose of study drug until disease progression, stable disease, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to 2 years)
  DCR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1 and mRECIST.
Duration of response (DOR) by RECIST 1.1 and mRECIST | From the first documentation of CR or PR to the first date of documentation of disease progression or death whichever occurs first (up to 2 years)
  DOR is defined as the time from the first documentation of CR or PR to the date of first documentation of disease progression or death (whichever occurs first) as assessed by RECIST 1.1 and mRECIST
Progression-free survival rate (PFSR) by RECIST 1.1 and mRECIST | From date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurs first (up to 2 years)
  PFSR in 6- and 12-months
Overall survival rate (OSR) | From date of first dose of study drug to the date of first documentation of death from any cause, whichever occurs first (up to 2 years)
  OSR in 6- and 12-months
Progression-free survival time (mPFS) | From date of first dose of study drug to the date of first documentation of disease progression (up to 2 years)
  The progression-free survival time (mPFS) defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1 and mRECIST.
Median overall survival time (mOS) | From the start date of the Treatment Phase until date of death from any cause (up to 2 years)
  OS is measured from the start date of the Treatment Phase (date of first study dose) until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date, whichever comes earlier.

OTHER OUTCOMES:
Treatment-related adverse events | From the start date of the Treatment Phase until date of death from any cause (up to 2 years)
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No